CLINICAL TRIAL: NCT07215000
Title: Cleansing Options in Outpatient Setting to Improve Tolerance (COOP SIT) Trial
Brief Title: Cleansing Options in Out-Patient Setting to Improve Tolerance (COOP SIT) Trial
Acronym: COOP SIT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Morehouse School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2282829
Record Dates: First submitted 2025-07-15; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer Screening; Bowel Cleansing for Colonoscopy
Keywords: Colorectal cancer screening; Bowel cleansing for colonoscopy
MeSH Terms: interventions — Golytely; polyethylene glycol 3350; Potassium Chloride; Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Golytely (Active Comparator): GoLYTELY is a prescription medicine used by adults to clean the colon before a colonoscopy or barium enema X-ray examination. GoLYTELY cleans your colon by causing you to have diarrhea (loose stools). Cleaning your colon helps your healthcare provider see the inside of your colon more clearly during your colonoscopy. Drink reconstituted solution at a rate of 8 ounces every 10 minutes, until 4 liters are consumed, or rectal effluent is clear.
  Interventions: Drug: Golytely
- Sulfave (Other): Suflave is a combination, osmotic prescription laxative that may be used to cleanse the bowel in preparation for colonoscopy in adults. Suflave contains polyethylene glycol 3350, sodium sulfate, potassium chloride, magnesium sulfate, and sodium chloride, and is supplied as a powder that is mixed with a low volume of water before consuming. It tastes like a lemon-lime sports drink. Drink 8 ounces of the solution every 15 minutes until the bottle is empty, and then drink an additional 16 ounces of water during the evening. One dose of Suflave is equal to one bottle plus one flavor-enhancing packet.
  Interventions: Drug: Sulfave
- Sutab (Other): SUTAB comes in a kit that contains two medication bottles and a cup for water. Each bottle contains 12 tablets (pills). You'll take 12 pills (one bottle) with water from the cup the night before your exam. Later that evening, drink two more cups of water. Fill the cup to the line each time. Then, six hours before your exam, repeat all three of those steps.
  Interventions: Drug: Sutab

INTERVENTIONS:
Drug: Golytely — large volume liquid prep.
  Arms: Golytely
Drug: Sulfave — SUFLAVE is a split-dose (2-day) regimen. A total of 2 bottles are required for complete preparation for colonoscopy. You will take 2 bottles of liquid in two separate doses. One dose of SUFLAVE is equal to one bottle plus one flavor enhancing packet.
  Other Names: polyethylene glycol 3350; sodium sulfaten; potassium chloride, magnesium sulfate
  Arms: Sulfave
Drug: Sutab — SUTAB comes in a kit that contains two medication bottles and a cup for water. Each bottle contains 12 tablets (pills). You'll take 12 pills (one bottle) with water from the cup the night before your exam. Later that evening, drink two more cups of water. Fill the cup to the line each time. Then, six hours before your exam, repeat all three of those steps.
  Arms: Sutab

SUMMARY:
The purpose of this research is to compare patient preferences for two bowel preparation options: low-volume tablets (Suflave/Sutab) versus the standard colon preparation using Golytely (polyethylene glycol). The study aims to enroll approximately 300 patients, who will be randomly assigned to one of the two preparation methods in a 2:1 ratio prior to their scheduled colonoscopy appointments. Surveys will be conducted both before and after the procedures.

This project will be conducted over a 12-month period and seeks to compare patient experience of both preparation methods in an outpatient setting. The study will evaluate the rate of preparation completion, patient satisfaction, tolerance of the solutions, and the endoscopic adequacy of each method.

Eligible participants are patients aged 18 or older with upcoming colonoscopy appointments who can provide informed consent in English or Spanish. There is no health risks associated with this study, as both bowel preparation methods are FDA-approved and commonly used in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age of 18 years undergoing outpatient colonoscopy for various indications, ability to consent in English or Spanish. Patients will still be allowed to join if there is a history of colorectal cancer or previous surgery

Exclusion Criteria:

* Patient is less than 18 years of age, any pregnant or nursing women, unable to consent, or patient is incarcerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Patient Experience | Until the end of the study
  Evaluate the patient experience of the two new colon prep options (low volume and tablets) versus conventional bowel prep in an out-patient setting.
Edoscopic Adequacy | Until the end of the study
  Assess endoscopic adequacy of the three bowel cleansing solutions

SECONDARY OUTCOMES:
Rate of Completion | Until the end of the study
  Determine the rate of completion for each colon prep option

OTHER OUTCOMES:
Rate of cancellation and patient satisfaction and tolerance | Until the end of the study
  Compare rate of cancelation/missed rate, patient satisfaction and tolerance for the three colon preps.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus M Luevano, MD, MS, Principal Investigator — Morehouse School of Medicine
Locations (1):
- Morehouse School of Medicine, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Averous M. [Results of early surgery of obstructive uropathies diagnosed prenatally: apropos of 56 cases]. Acta Urol Belg. 1989;57(2):423-30. No abstract available. French. PMID 2763922
- [Background] Niikawa N, Ishikiriyama S, Shikimani T. The "Michelin tire baby" syndrome--an autosomal dominant trait. Am J Med Genet. 1985 Nov;22(3):637-8. doi: 10.1002/ajmg.1320220327. No abstract available. PMID 4061498
- [Background] Ito F, Harada Y. Responses of muscle spindle and leaflike receptor afferents to sinusoidal stretching. Am J Physiol. 1972 Nov;223(5):1246-9. doi: 10.1152/ajplegacy.1972.223.5.1246. No abstract available. PMID 4265954
- [Background] Adamski GB, Garin EH, Ballinger WE, Shulman ST. Generalized nonsuppurative myositis with staphylococcal septicemia. J Pediatr. 1980 Apr;96(4):694-7. doi: 10.1016/s0022-3476(80)80745-1. No abstract available. PMID 7359276
- [Background] Jaric MV. Long-range icosahedral orientational order and quasicrystals. Phys Rev Lett. 1985 Aug 5;55(6):607-610. doi: 10.1103/PhysRevLett.55.607. No abstract available. PMID 10032399
- [Background] Vemulapalli KC, Lahr RE, Rex DK. 2021 Patient Perceptions Regarding Colonoscopy Experience. J Clin Gastroenterol. 2023 Apr 1;57(4):400-403. doi: 10.1097/MCG.0000000000001689. PMID 35324481
- [Background] Chien C, Morimoto LM, Tom J, Li CI. Differences in colorectal carcinoma stage and survival by race and ethnicity. Cancer. 2005 Aug 1;104(3):629-39. doi: 10.1002/cncr.21204. PMID 15983985
- [Background] Miller JS, Cervenka T, Lund J, Okazaki IJ, Moss J. Purine metabolites suppress proliferation of human NK cells through a lineage-specific purine receptor. J Immunol. 1999 Jun 15;162(12):7376-82. PMID 10358189
- [Background] Wilson NI, Dreghorn CR. Costs of prophylaxis in joint prosthesis. Br Med J (Clin Res Ed). 1988 Feb 13;296(6620):499. No abstract available. PMID 3126877
- [Background] Freer JH, Levinson HS. Fine structure of Bacillus megaterium during microcycle sporogenesis. J Bacteriol. 1967 Aug;94(2):441-57. doi: 10.1128/jb.94.2.441-457.1967. PMID 4962705
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525